CLINICAL TRIAL: NCT02951780
Title: A Randomized, 9-Way, Single-Dose, Crossover Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of LY3185643 and rGlucagon in Healthy Subjects
Brief Title: A Study of LY3185643 and rGlucagon in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16502; I8Z-MC-APCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3185643 (Experimental): LY3185643 administered subcutaneous (SC)
  Interventions: Drug: LY3185643
- rGlucagon (Experimental): rGlucagon administered subcutaneous (SC)
  Interventions: Drug: rGlucagon

INTERVENTIONS:
Drug: LY3185643 — Administered SC
  Arms: LY3185643
Drug: rGlucagon — Administered SC
  Arms: rGlucagon

SUMMARY:
The purpose of this study is to determine how the body handles LY3185643 and rGlucagon and what effects LY3185643 and rGlucagon have on the body. This study will also help to determine if LY3185643 is safe and well-tolerated.

This study will last at least 35 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical history and physical examination
* Body mass index of 18.0 to 30.0 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Have participated, within the last 30 days, in a clinical trial involving an investigational product
* Known allergies to LY3185643 or rGlucagon, related compounds, or any components of the formulation
* History or electrocardiogram (ECG) evidence of heart block, or any abnormality in the 12-lead ECG
* Abnormal blood pressure
* History of recurring symptomatic postural hypotension irrespective of the decrease in blood pressure, or asymptomatic postural hypotension at screening as defined as a decrease in systolic blood pressure greater than or equal to (≥) 20 millimeter of Mercury (mm Hg) within 3 minutes when changing from supine to standing position
* History of vasovagal response such as fainting
* History of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* History of/current insulinoma and/or pheochromocytoma
* Have used systemic glucocorticoids within 3 months before entry into the study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com. This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study with three periods. Each participant received up to 3 doses of study drug (rGlucagon and/or LY3185643) in a dosing day as per the dosing sequence in each period with 7 to 12 days washout period.
Groups:
- Cohort A (Sequence 1-9-7: 6-4-8: 5-3-2): LY3185643 and rGlucagon were administered as single subcutaneous (SC) doses with Dosing Sequence 1-9-7 in Treatment Period 1, Dosing Sequence: 6-4-8 in Treatment Period 2 and Dosing Sequence: 5-3-2 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 microgram (μg) LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort B (Sequence 2,7,8: 4,5,9: 6,1,3 ): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 2-7-8 in Treatment Period 1, Dosing Sequence: 4-5-9 in Treatment Period 2 and Dosing Sequence: 6-1-3 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort C (Sequence 3,8,9: 5,6,7: 4,2,1): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 3-8-9 in Treatment Period 1, Dosing Sequence: 5-6-7 in Treatment Period 2 and Dosing Sequence: 4-2-1 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort D (Sequence 4,6,2: 3,9,1: 8,7,5): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 4-6-2 in Treatment Period 1, Dosing Sequence: 3-9-1 in Treatment Period 2 and Dosing Sequence: 8-7-5 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort E (Sequence 5,4,3: 1,7,2: 9,8,6): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 5-4-3 in Treatment Period 1, Dosing Sequence: 1-7-2 in Treatment Period 2 and Dosing Sequence: 9-8-6 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort F (Sequence 6,5,1: 2,8,3: 7,9,4): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 6-5-1 in Treatment Period 1, Dosing Sequence: 2-8-3 in Treatment Period 2 and Dosing Sequence: 7-9-4 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort G (Sequence 7,1,4: 9,2,6: 9,2,6): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 7-1-4 in Treatment Period 1, Dosing Sequence: 9-2-6 in Treatment Period 2 and Dosing Sequence: 9-2-6 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort H (Sequence 8,2,5: 7,3,4: 1,6,9): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 8-2-5 in Treatment Period 1, Dosing Sequence: 7-3-4 in Treatment Period 2 and Dosing Sequence: 1-6-9 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Cohort I (Sequence 9,3,6: 8,1,5: 2,4,7) ): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 9-3-6 in Treatment Period 1, Dosing Sequence: 8-1-5 in Treatment Period 2 and Dosing Sequence: 2-4-7 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
Period: Period 1
Arm/Group | Cohort A (Sequence 1-9-7: 6-4-8: 5-3-2) | Cohort B (Sequence 2,7,8: 4,5,9: 6,1,3 ) | Cohort C (Sequence 3,8,9: 5,6,7: 4,2,1) | Cohort D (Sequence 4,6,2: 3,9,1: 8,7,5) | Cohort E (Sequence 5,4,3: 1,7,2: 9,8,6) | Cohort F (Sequence 6,5,1: 2,8,3: 7,9,4) | Cohort G (Sequence 7,1,4: 9,2,6: 9,2,6) | Cohort H (Sequence 8,2,5: 7,3,4: 1,6,9) | Cohort I (Sequence 9,3,6: 8,1,5: 2,4,7) )
Started | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 2
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Scheduling Conflicts | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Cohort A (Sequence 1-9-7: 6-4-8: 5-3-2) | Cohort B (Sequence 2,7,8: 4,5,9: 6,1,3 ) | Cohort C (Sequence 3,8,9: 5,6,7: 4,2,1) | Cohort D (Sequence 4,6,2: 3,9,1: 8,7,5) | Cohort E (Sequence 5,4,3: 1,7,2: 9,8,6) | Cohort F (Sequence 6,5,1: 2,8,3: 7,9,4) | Cohort G (Sequence 7,1,4: 9,2,6: 9,2,6) | Cohort H (Sequence 8,2,5: 7,3,4: 1,6,9) | Cohort I (Sequence 9,3,6: 8,1,5: 2,4,7) )
Started | 3 | 2 | 3 | 2 | 2 | 3 | 2 | 2 | 2
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 2 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Scheduling Conflicts | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Cohort A (Sequence 1-9-7: 6-4-8: 5-3-2) | Cohort B (Sequence 2,7,8: 4,5,9: 6,1,3 ) | Cohort C (Sequence 3,8,9: 5,6,7: 4,2,1) | Cohort D (Sequence 4,6,2: 3,9,1: 8,7,5) | Cohort E (Sequence 5,4,3: 1,7,2: 9,8,6) | Cohort F (Sequence 6,5,1: 2,8,3: 7,9,4) | Cohort G (Sequence 7,1,4: 9,2,6: 9,2,6) | Cohort H (Sequence 8,2,5: 7,3,4: 1,6,9) | Cohort I (Sequence 9,3,6: 8,1,5: 2,4,7) )
Started | 3 | 2 | 3 | 2 | 2 | 3 | 2 | 1 | 2
Completed | 3 | 2 | 3 | 2 | 2 | 3 | 2 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Cohort A (Sequence 1,9,7: 6,4,8:5,3,2): LY3185643 and rGlucagon were administered as single SC doses with Dosing Sequence 1-9-7 in Treatment Period 1, Dosing Sequence: 6-4-8 in Treatment Period 2 and Dosing Sequence: 5-3-2 in Treatment Period 3.
  Dose assignment was: Dose 1 = 10 μg LY3185643; Dose 2 = 25 μg LY3185643; Dose 3 = 50 μg LY3185643; Dose 4 = 100 μg LY3185643; Dose 5 = 200 μg LY3185643; Dose 6 = 10 μg rGlucagon; Dose 7 = 25 μg rGlucagon; Dose 8 = 50 μg rGlucagon; Dose 9 = 200 μg rGlucagon.
- Total: Total of all reporting groups
Arm/Group | Cohort A (Sequence 1,9,7: 6,4,8:5,3,2) | Cohort B (Sequence 2,7,8: 4,5,9: 6,1,3 ) | Cohort C (Sequence 3,8,9: 5,6,7: 4,2,1) | Cohort D (Sequence 4,6,2: 3,9,1: 8,7,5) | Cohort E (Sequence 5,4,3: 1,7,2: 9,8,6) | Cohort F (Sequence 6,5,1: 2,8,3: 7,9,4) | Cohort G (Sequence 7,1,4: 9,2,6: 9,2,6) | Cohort H (Sequence 8,2,5: 7,3,4: 1,6,9) | Cohort I (Sequence 9,3,6: 8,1,5: 2,4,7) ) | Total
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 2 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 2 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 2 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 2 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 2 | 23

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of LY3185643 and rGlucagon
Description: Maximum observed plasma concentration (Cmax) was assessed for LY3185643 and rGlucagon.
Time Frame: 0 (pre-dose), 15, 30, 60, 120 and 180 minutes post-dose
Population: All randomized participants who received at least one dose of study drug (LY3185643, rGlucagon) and with a baseline and at least 1 postbaseline measurement for each dose with evaluable LY3185643 and rGlucagon PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Groups:
- 10 ug LY3185643: LY3185643 has been administered SC as single dose of 10 ug.
- 25 ug LY3185643: LY3185643 has been administered SC as single dose of 25 ug.
- 50 ug LY3185643: LY3185643 has been administered SC as single dose of 50 ug.
- 100 ug LY3185643: LY3185643 has been administered SC as single dose of 100 ug.
- 200 ug LY3185643: LY3185643 has been administered SC as single dose of 200 ug.
- 10 ug rGlucagon: rGlucagon has been administered SC as single dose of 10 ug.
- 25 ug rGlucagon: rGlucagon has been administered SC as single dose of 25 ug.
- 50 ug rGlucagon: rGlucagon has been administered SC as single dose of 50 ug.
- 200 ug rGlucagon: rGlucagon has been administered SC as single dose of 200 ug.
Arm/Group | 10 ug LY3185643 | 25 ug LY3185643 | 50 ug LY3185643 | 100 ug LY3185643 | 200 ug LY3185643 | 10 ug rGlucagon | 25 ug rGlucagon | 50 ug rGlucagon | 200 ug rGlucagon
Number analyzed (Participants) | 19 | 22 | 20 | 21 | 21 | 19 | 21 | 22 | 20
picogram per milliliter (pg/mL) | 191 (49) | 658 (36) | 1110 (40) | 2010 (40) | 3830 (38) | 53.7 (31) | 204 (70) | 283 (44) | 897 (49)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3185643 and rGlucagon
Description: Area under the concentration versus time curve from zero to infinity (AUC0-inf) was assessed for LY3185643 and rGlucagon.
Time Frame: 0 (pre-dose), 15, 30, 60, 120 and 180 minutes post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour per milliliter (pg*hr/mL)
Arm/Group | 10 ug LY3185643 | 25 ug LY3185643 | 50 ug LY3185643 | 100 ug LY3185643 | 200 ug LY3185643 | 10 ug rGlucagon | 25 ug rGlucagon | 50 ug rGlucagon | 200 ug rGlucagon
Number analyzed (Participants) | 4 | 20 | 19 | 18 | 15 | 19 | 15 | 20 | 20
picogram*hour per milliliter (pg*hr/mL) | 356 (30) | 1200 (21) | 2230 (21) | 4430 (21) | 9120 (17) | NA (NA) — AUC(0-inf) could not be calculated because of several PK samples were below the quantification limit. | 189 (57) | 249 (24) | 764 (26)

3. Primary Outcome: Pharmacodynamics (PD): Change From Baseline in Maximum Concentration (Cmax) of Blood Glucose of LY3185643 and rGlucagon
Description: Cmax was assessed for LY3185643 and rGlucagon.
Time Frame: -5, 0 (pre-dose), 5, 10, 15, 22, 30, 45, 60, 75, 90, 105, 120, 150, 180 minutes post-dose
Population: All randomized participants who received at least one dose of study drug (LY3185643, rGlucagon) and with a baseline and at least 1 postbaseline measurement for each dose with evaluable LY3185643 and rGlucagon PD data.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | 10 ug LY3185643 | 25 ug LY3185643 | 50 ug LY3185643 | 100 ug LY3185643 | 200 ug LY3185643 | 10 ug rGlucagon | 25 ug rGlucagon | 50 ug rGlucagon | 200 ug rGlucagon
Number analyzed (Participants) | 20 | 23 | 21 | 22 | 22 | 21 | 21 | 22 | 20
milligram per deciliter (mg/dL) | 5.54 (2.66) | 15.1 (9.94) | 24.0 (16.6) | 37.1 (20.6) | 53.2 (17.7) | 4.37 (3.39) | 12.5 (11.1) | 16.9 (11.4) | 38.1 (13.9)

4. Primary Outcome: Pharmacodynamics (PD): Change From Baseline in Maximum Concentration (Cmax) of C-peptide of LY3185643 and rGlucagon
Description: Cmax was assessed for C-peptide of LY3185643 and rGlucagon
Time Frame: -5, 0 (predose), 5, 15, 30, 60 and 120 minutes post-dose
Population: All randomized participants who received at least one dose of study drug (C-peptide of LY3185643 and rGlucagon) and with a baseline and at least 1 postbaseline measurement for each dose with evaluable LY3185643 and rGlucagon PD data.
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | 10 ug LY3185643 | 25 ug LY3185643 | 50 ug LY3185643 | 100 ug LY3185643 | 200 ug LY3185643 | 10 ug rGlucagon | 25 ug rGlucagon | 50 ug rGlucagon | 200 ug rGlucagon
Number analyzed (Participants) | 20 | 23 | 21 | 22 | 22 | 21 | 21 | 22 | 20
picomole per liter (pmol/L) | 50.2 (44.7) | 201 (168) | 324 (330) | 555 (387) | 969 (451) | 25.4 (34.1) | 119 (98.9) | 218 (154) | 577 (292)

5. Primary Outcome: Pharmacodynamics (PD): Change From Baseline in Area Under the Concentration Time Curve (AUC) of Blood Glucose of LY3185643 and rGlucagon
Description: Area under the concentration versus time curve from time zero to 3 hours [AUC (0-3)] was assessed for LY3185643 and rGlucagon.
Time Frame: -5, 0 (pre-dose), 5, 10, 15, 22, 30, 45, 60, 75, 90, 105, 120, 150, 180 minutes post-dose
Population: All randomized participants who received at least one dose of study drug (LY3185643, C-peptide) and with a baseline and at least 1 postbaseline measurement for each dose with evaluable LY3185643 and rGlucagon PD data.
Measure: Mean (Standard Deviation); unit: milligram*hour per deciliter (mg*hr/dL)
Arm/Group | 10 ug LY3185643 | 25 ug LY3185643 | 50 ug LY3185643 | 100 ug LY3185643 | 200 ug LY3185643 | 10 ug rGlucagon | 25 ug rGlucagon | 50 ug rGlucagon | 200 ug rGlucagon
Number analyzed (Participants) | 20 | 23 | 21 | 22 | 22 | 21 | 21 | 22 | 20
milligram*hour per deciliter (mg*hr/dL) | 1.46 (7.52) | 18.9 (15.3) | 29.7 (21.1) | 45.1 (27.1) | 71.5 (37.8) | 0.594 (11.9) | 7.74 (15.6) | 12.1 (14.4) | 24.0 (15.8)

6. Primary Outcome: Pharmacodynamics (PD): Change From Baseline in Area Under the Concentration Time Curve (AUC) of C-Peptide of LY3185643 and rGlucagon
Description: Area under the concentration versus time curve from time zero to 3 hours [AUC (0-3)] was assessed for C-peptide of LY3185643 and rGlucagon.
Time Frame: -5, 0 (pre-dose), 5, 15, 30, 60 and 120 minutes post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: picomole*hour per liter (pmol*h/L)
Arm/Group | 10 ug LY3185643 | 25 ug LY3185643 | 50 ug LY3185643 | 100 ug LY3185643 | 200 ug LY3185643 | 10 ug rGlucagon | 25 ug rGlucagon | 50 ug rGlucagon | 200 ug rGlucagon
Number analyzed (Participants) | 20 | 23 | 21 | 22 | 22 | 21 | 21 | 22 | 20
picomole*hour per liter (pmol*h/L) | 25.0 (60.5) | 246 (194) | 354 (388) | 669 (441) | 1170 (529) | -28.3 (82.2) | 82.1 (130) | 167 (162) | 626 (325)

ADVERSE EVENTS:
Time Frame: Up To 3 Months
Description: All randomized participants who received at least one dose of study drug (LY3185643, rGlucagon).
Arm/Group | 10 ug LY3185643 | 25 ug LY3185643 | 50 ug LY3185643 | 100 ug LY3185643 | 200 ug LY3185643 | 10 ug rGlucagon | 25 ug rGlucagon | 50 ug rGlucagon | 200 ug rGlucagon
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23 | 0/21 | 0/22 | 0/22 | 0/21 | 0/21 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23 | 0/21 | 0/22 | 0/22 | 0/21 | 0/21 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 3/23 | 3/21 | 5/22 | 4/22 | 2/21 | 1/21 | 2/22 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 ug LY3185643 (N=20) | 25 ug LY3185643 (N=23) | 50 ug LY3185643 (N=21) | 100 ug LY3185643 (N=22) | 200 ug LY3185643 (N=22) | 10 ug rGlucagon (N=21) | 25 ug rGlucagon (N=21) | 50 ug rGlucagon (N=22) | 200 ug rGlucagon (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT02951780/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT02951780/SAP_001.pdf